CLINICAL TRIAL: NCT00224068
Title: A Multicenter, Randomized, Controlled Prospective Trial of the Safety and Efficacy of Ferrlecit® in Anemic Cancer Patients Who Are Receiving Acute Chemotherapy and Epoetin as Compared to Oral Iron and No Treatment
Brief Title: Effect of Iron Therapy as an Adjunct to Epoetin Alfa in the Anemia of Cancer Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR01008
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Anemia
Keywords: Iron deficiency; Sodium ferric gluconate; anemia; cancer chemotherapy; epoetin alfa; Anemia/drug therapy; Anemia, Iron-Deficiency/drug therapy/etiology; Hematinics/administration & dosage/pharmacology; Antineoplastic Agents/adverse effects; Erythropoietin, Recombinant/therapeutic use/adverse effects
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — ferric gluconate; ferrous sulfate; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sodium ferric gluconate, ferrous sulfate, standard of care

SUMMARY:
This study evaluates the safety and efficacy of Ferrlecit® (ferric gluconate; a form of intravenous iron) or ferrous sulfate (a form of oral iron) in improving the response to epoetin alfa among anemic cancer patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonmyeloid malignancy
* Moderate to severe anemia
* Adequate iron stores as measured by either TSAT or ferritin
* About to start cycle of chemotherapy
* Eligible for epoetin alfa therapy

Exclusion Criteria:

* Highly elevated TSAT or ferritin
* Recent transfusion, epoetin alfa, darbepoetin or intravenous iron
* Medical conditions that would confound the efficacy evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2002-05; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin

SECONDARY OUTCOMES:
Change in various iron indices

CONTACTS AND LOCATIONS:
Overall Officials: Naomi V. Dahl, Pharm.D., Study Director — Watson Laboratories, Inc.
Locations (32):
- United States (32):
  - Bakersfield, California
  - Chula Vista, California
  - Long Beach, California
  - Los Angeles, California
  - Norwich, Connecticut
  - Port Saint Lucie, Florida
  - Zephyrhills, Florida
  - Columbus, Georgia
  - Coeur d'Alene, Idaho
  - Hutchinson, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Saint Joseph, Michigan
  - Southfield, Michigan
  - Duluth, Minnesota
  - Greenwood, Mississippi
  - Cherry Hill, New Jersey
  - Denville, New Jersey
  - Manhasset, New York
  - Bismarck, North Dakota
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Chester, Pennsylvania
  - Columbia, South Carolina
  - Laredo, Texas
  - Richmond, Virginia
  - Salem, Virginia
  - Walla Walla, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Henry DH, Dahl NV, Auerbach M, Tchekmedyian S, Laufman LR. Intravenous ferric gluconate significantly improves response to epoetin alfa versus oral iron or no iron in anemic patients with cancer receiving chemotherapy. Oncologist. 2007 Feb;12(2):231-42. doi: 10.1634/theoncologist.12-2-231. PMID 17296819